CLINICAL TRIAL: NCT05650606
Title: Inpatient Rehabilitation and Post-Discharge Outcomes of Patients With Stroke Participating in High Intensity Gait Training
Brief Title: Inpatient Rehabilitation and Post-Discharge Outcomes With High Intensity Gait Training (HIGT) of Patients With Stroke
Acronym: HIGT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Sunnyview Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Patricia Broschart Valenza, Therapy Supervisor, Sunnyview Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0912-1
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Vascular Accident
Keywords: High Intensity Gait Training; Inpatient Rehabilitation; Health Care Burden
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Gait Training (Experimental): HIGT will be performed 4-6 times per week in place of conventional physical therapy. The patient's heart rate(HR)and blood pressure(BP) will be measured throughout each session. If the HR or BP is out of the acceptable range, patients will undergo standard physical therapy for that session, and the medical team will be contacted.
  Target HR zones will be calculated with the Karvonen formula. The first session goal is to reach a target HR range that is 50-60% of heart rate reserve. The goal for subsequent sessions is to reach 70-80% of heart rate reserve. Rate of perceived exertion (RPE) will also be utilized.
  The primary therapist will design an individualized HIGT treatment program with a combination of speed dependent treadmill activities, activity-based treadmill activities, stair training, and over ground activities.
  The patient will be reminded during each session to ask for a rest as needed. Standing rests are preferred over sitting rests, but either may be utilized.
  Interventions: Other: High Intensity Gait Training
- Conventional (Active Comparator): The conventional physical therapy sessions are what a patient would normally receive during their rehabilitation. Physical therapy sessions are usually 60-90 minutes per day for 5 days each week, and possibly one 30-minute session on a 6th day. Physical therapy sessions are focused on gait, balance, and strengthening activities to address goals related to functional mobility. Clinicians administering therapy to patients in this arm will not be given instructions on the types of therapies they administer; however, they will not be permitted to do HIGT with patients. Therapists will be permitted to use other devices such as Ekso exoskeleton, Lite Gait, Rifton Tram Body Weight Support Devices, and Electrical Stimulation devices including the XCITE and RT300.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: High Intensity Gait Training — Physical therapy intervention for improving gait in patients post Cerebral Vascular Accident.
  Arms: High Intensity Gait Training
Other: Conventional Therapy — Standard inpatient rehabilitation physical therapy treatments for Cerebral Vascular Accident.
  Arms: Conventional

SUMMARY:
Stroke is a major cause of disability, with 2-3% of Americans reporting stroke related impairments (Tsao 2022). Following stroke, over half of Medicare patients are discharged to post-acute care facilities or receive home-based health care (Tsao 2022). Inpatient rehabilitation guidelines are lacking, with many interventions based on research of patients with chronic stroke. There is great need for randomized clinical trials during the early subacute period (Bernhardt 2017, Jordan 2021).

Clinical practice guidelines recommend high intensity gait training (HIGT) for ambulatory patients with chronic stroke (Hornby 2020). Outpatient HIGT protocols incorporating variable stepping demonstrate equivalent effectiveness to forward stepping protocols (Hornby 2019) and have yielded superior results to lower intensity therapies (Hornby 2019, Hornby 2016). Research suggests that HIGT with variable stepping is feasible during inpatient rehabilitation (Hornby 2015, Moore 2020). Pre-post studies suggest that participation in HIGT during inpatient rehabilitation yields greater improvements in walking without an increase in adverse events. (Moore 2020). Despite this, there are no randomized controlled trials evaluating HIGT in the inpatient setting.

The subacute phase of stroke recovery may be a critical time for neuroplasticity (Dromerick 2021). Not only might rehabilitation interventions be more effective when initiated earlier (Biernaskie 2004, Dromerick 2021) but because inpatient rehabilitation represents the transition from hospital to home, interventions during this timeframe have the potential to improve discharge disposition, enhance quality of life, and reduce utilization of post-discharge services.

In this randomized controlled study, investigators will determine how participation in HIGT during inpatient rehabilitation affects balance, ambulation, and quality of life after 14 and/or 21 days of inpatient rehabilitation, and 8 weeks post-discharge. Investigators will also determine if HIGT reduces health care burden with a cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* adults (≥18 years) recovering from a unilateral cerebral infarct with resultant hemiparesis occurring less than three months prior. Patients must have an expected length of stay of at least 14 days.

Exclusion Criteria:

* are older than 85 years of age have evidence of intracranial hemorrhage on head imaging

  * have had a brainstem, cerebellar or bilateral hemisphere stroke
  * are medically unstable
  * are pregnant
  * have chronic cardiorespiratory disease

    * on oxygen
    * angina
    * unstable arrhythmias
    * ischemic cardiomyopathy (Ejection Fraction <50%)
  * unable to follow 2 steps commands accurately
  * neurological comorbidities that affect gait

    * Parkinson's
    * severe polyneuropathy
  * unable to walk at least 150 feet premorbid
  * dependent assistance level for transfer from a chair to a bed as assessed by physical therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
10 Meter Walk Test at Self Selected Speed | (Day 13-15) - (Day 1-3)
  Used to assess walking speed over a short distance at the patient's chosen speed.
10 Meter Walk Test at Self Selected Speed | (Day 20-22)- (Day 1-3)
  Used to assess walking speed over a short distance at the patient's chosen speed.
10 Meter Walk Test at Self Selected Speed | (Day 62 to Day 86)-(Day 14 to Day 21)
  Used to assess walking speed over a short distance at the patient's chosen speed.
10 Meter Walk Test at Fast Speed | (Day 13-15) - (Day 1-3)
  Used to assess walking speed over a short distance at the patient's self determined speed that is as fast as they can safely walk..
10 Meter Walk Test at Fast Speed | (Day 20-22) - (Day 1-3)
  Used to assess walking speed over a short distance at the patient's self determined speed that is as fast as they can safely walk..
10 Meter Walk Test at Fast Speed | (Day 62 to Day 86)-(Day 14 to Day 21)
  Used to assess walking speed over a short distance at the patient's self determined speed that is as fast as they can safely walk..
6 Minute Walk Test | (Day 13-15) - (Day 1-3)
  Used to assess walking endurance and aerobic capacity. The total distance the patient walks over six minutes is recorded.
6 Minute Walk Test | (Day 20-22) - (Day 1-3)
  Used to assess walking endurance and aerobic capacity. The total distance the patient walks over six minutes is recorded.
6 Minute Walk Test | (Day 62 to Day 86)-(Day 14 to Day 21)
  Used to assess walking endurance and aerobic capacity. The total distance the patient walks over six minutes is recorded.
Stroke Impact Scale (SIS) | (Day 62 to Day 86)-(Day 14 to Day 21)
  The Stroke Impact Scale (SIS) is a self report questionnaire that uses 9 categories to assess disability and quality of life after having had a stroke.
Life Space Assessment (LSA) | (Day 62 to Day 86)-(Day 14 to Day 21)
  The LSA is a self report tool that measures frequency of independent mobility using 9 questions.
Cost of inpatient rehabilitation and post-discharge health care services | (Day 62 to Day 86) - (Day 1 to Day 3)
  This will include the cost of home health care, outpatient therapies, subacute nursing facility and hospital readmissions

SECONDARY OUTCOMES:
BERG Balance Scale | (Day 13-15) - (Day 1-3)
  A 14 item scale used to assess sitting, standing, static and dynamic balance.
BERG Balance Scale | (Day 20-22) - (Day 1-3)
  A 14 item scale used to assess sitting, standing, static and dynamic balance.
BERG Balance Scale | (Day 62 to Day 86)-(Day 14 to Day 21)
  A 14 item scale used to assess sitting, standing, static and dynamic balance.
5 Times Sit to Stand | (Day 13-15) - (Day 1-3)
  Measures functional lower extremity strength and movement patterns used to complete functional movements
5 Times Sit to Stand | (Day 20-22) - (Day 1-3)
  Measures functional lower extremity strength and movement patterns used to complete functional movements
5 Times Sit to Stand | (Day 62 to Day 86)-(Day 14 to Day 21)
  Measures functional lower extremity strength and movement patterns used to complete functional movements
Functional Ambulation Category (FAC) | (Day 13-15) - (Day 1-3)
  A five point scale used to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
Functional Ambulation Category (FAC) | (Day 20-22) - (Day 1-3)
  A five point scale used to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
Functional Ambulation Category (FAC) | (Day 62 to Day 86)-(Day 14 to Day 21)
  A five point scale used to categorize a patient's ambulation status, ranging from independent walking outside to non-functional walking.
Assistive Device Use | (Day 13-15) - (Day 1-3)
  Document which (if any) assistive device the patient uses for ambulation.
Assistive Device Use | (Day 20-22) - (Day 1-3)
  Document which (if any) assistive device the patient uses for ambulation.
Assistive Device Use | (Day 62 to Day 86)-(Day 14 to Day 21)
  Document which (if any) assistive device the patient uses for ambulation.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Broschart Valenza, DPT, Principal Investigator — Sunnyview Rehabilitation Hospital
Locations (1):
- Sunnyview Rehabilitation Hospital, Schenectady, New York, United States

REFERENCES:
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed Definitions and a Shared Vision for New Standards in Stroke Recovery Research: The Stroke Recovery and Rehabilitation Roundtable Taskforce. Neurorehabil Neural Repair. 2017 Sep;31(9):793-799. doi: 10.1177/1545968317732668. PMID 28934920
- [Background] Biernaskie J, Chernenko G, Corbett D. Efficacy of rehabilitative experience declines with time after focal ischemic brain injury. J Neurosci. 2004 Feb 4;24(5):1245-54. doi: 10.1523/JNEUROSCI.3834-03.2004. PMID 14762143
- [Background] Dromerick AW, Geed S, Barth J, Brady K, Giannetti ML, Mitchell A, Edwardson MA, Tan MT, Zhou Y, Newport EL, Edwards DF. Critical Period After Stroke Study (CPASS): A phase II clinical trial testing an optimal time for motor recovery after stroke in humans. Proc Natl Acad Sci U S A. 2021 Sep 28;118(39):e2026676118. doi: 10.1073/pnas.2026676118. PMID 34544853
- [Background] Hornby TG, Holleran CL, Leddy AL, Hennessy P, Leech KA, Connolly M, Moore JL, Straube D, Lovell L, Roth E. Feasibility of Focused Stepping Practice During Inpatient Rehabilitation Poststroke and Potential Contributions to Mobility Outcomes. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):923-32. doi: 10.1177/1545968315572390. Epub 2015 Feb 26. PMID 25721233
- [Background] Hornby TG, Holleran CL, Hennessy PW, Leddy AL, Connolly M, Camardo J, Woodward J, Mahtani G, Lovell L, Roth EJ. Variable Intensive Early Walking Poststroke (VIEWS): A Randomized Controlled Trial. Neurorehabil Neural Repair. 2016 Jun;30(5):440-50. doi: 10.1177/1545968315604396. Epub 2015 Sep 3. PMID 26338433
- [Background] Hornby TG, Henderson CE, Plawecki A, Lucas E, Lotter J, Holthus M, Brazg G, Fahey M, Woodward J, Ardestani M, Roth EJ. Contributions of Stepping Intensity and Variability to Mobility in Individuals Poststroke. Stroke. 2019 Sep;50(9):2492-2499. doi: 10.1161/STROKEAHA.119.026254. Epub 2019 Aug 22. PMID 31434543
- [Background] Hornby TG, Reisman DS, Ward IG, Scheets PL, Miller A, Haddad D, Fox EJ, Fritz NE, Hawkins K, Henderson CE, Hendron KL, Holleran CL, Lynskey JE, Walter A; and the Locomotor CPG Appraisal Team. Clinical Practice Guideline to Improve Locomotor Function Following Chronic Stroke, Incomplete Spinal Cord Injury, and Brain Injury. J Neurol Phys Ther. 2020 Jan;44(1):49-100. doi: 10.1097/NPT.0000000000000303. PMID 31834165
- [Background] Jordan N, Deutsch A. (2021). Why and How to Demonstrate the Value of Rehabilitation Services. ACRM, 000:1-6. https://doi.org/10.1016/j.apmr.2021.06.028
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Moore JL, Nordvik JE, Erichsen A, Rosseland I, Bo E, Hornby TG; FIRST-Oslo Team. Implementation of High-Intensity Stepping Training During Inpatient Stroke Rehabilitation Improves Functional Outcomes. Stroke. 2020 Feb;51(2):563-570. doi: 10.1161/STROKEAHA.119.027450. Epub 2019 Dec 30. PMID 31884902